CLINICAL TRIAL: NCT02101671
Title: Inadequate Emergence After Anaesthesia in Laparoscopic Surgery in Trendelemburg Position
Brief Title: Inadequate Emergence After Laparoscopic Surgery in Trendelemburg Position
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Morena Basso, MD, Corporacion Parc Tauli
Other Study IDs: 2014/522
Record Dates: First submitted 2014-03-29; First posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Delayed Emergence From Anesthesia; Delirium, Cause Unknown; Confusion; Disorientation on Emergence
Keywords: agitation; anaesthesia; laparoscopy; surgery; delirium; sedation; emergence; steep; trendelemburg; position; delayed; Confusion; Disorientation
MeSH Terms: conditions — Delayed Emergence from Anesthesia; Delirium; Confusion; Psychomotor Agitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- trendelemburg positioning: Patients undergone laparoscopic surgery in trendelemburg position
- Not trendelemburg positioning: Patients undergone laparoscopic surgery not in trendelemburg position

SUMMARY:
The purpose of this study is to determinate if the patients submitted to laparoscopic surgery in trendelemburg position develope more inadequate anaesthesic emergence than patients submitted to laparoscopic surgery in other positions.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic surgery
* general anaesthesia
* trendelemburg positioning
* extubated in the operatory theater

Exclusion Criteria:

* unable of communicate
* dementia
* psychiatric history
* neurosurgery
* alchohol and drugs addictions

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient undergone surgery
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-08 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Inadequate emergence after anaesthesia | 10 minutes after the arrival of the patient in the postsurgical unit
  The inadequate emergence after anaesthesia will be evalueted with the Richmond Agitation Sedation Scale, defining as inadequate emergence a punctuation >= +1 (delirium form) and <=-2 (hypoactive form).

CONTACTS AND LOCATIONS:
Overall Officials: Morena Basso, Principal Investigator — Corporacion Parc Tauli
Locations (1):
- Anaesthesia and Reanimation Department, Hospital Parc Tauli, Sabadell, Barcelona, Spain